CLINICAL TRIAL: NCT03585933
Title: Prognostic Value of Myocardial Fibrosis in Severe Aortic Valve Stenosis
Acronym: FIB-AS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Peter Sogaard,MD DMSc, Peter Sogaard, Clinical Professor, Vilnius University
Other Study IDs: 1014; 09.3.3-LMT-K-712 (Other Grant/Funding Number: European structural funds)
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Aortic Stenosis, Calcific
Keywords: Myocardial fibrosis; Severe aortic stenosis; Cardiovascular magnetic resonance; Scintigraphy; SAVR/TAVI
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum, myocardial tissue samples obtained intra-operatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging — Echocardiography: assessment of aortic stenosis severity, evaluation of LV diastolic and systolic function; CMR: chambers quantification, LGE, T1 mapping; Intraoperative myocardial tissue biopsy for patients undergoing SAVR; DPD scintigraphy: assessment of cardiac transthyretin amyloidosis
  Other Names: echocardiography; Intra-operative myocardial biopsy

SUMMARY:
Degenerative aortic valve stenosis (AS) is the most common valve heart disease in the developed Western countries. The hemodynamic progression of AS occurs over time and leads to LV hypertrophy (LVH) as a compensation mechanism of the heart. Morphological changes such as increasing muscle fibre thickness, collagen volume, and interstitial fibrosis occur in AS patients. These changes result in left ventricular (LV) diastolic and systolic dysfunction and, consequently, to with AS related symptoms. When symptoms associated with AS appear, patients' prognosis is poor if surgical aortic valve replacement (SAVR) or a trans-catheter aortic valve implantation (TAVI) is not performed.

Primary hypothesis of the research: fibrotic changes in the myocardium are related to immediate (in hospital) or long-term complications (MACE and all-cause mortality) in patients with severe AS.

The goal of the study is to determine the prognostic implications of focal as well as diffuse myocardial fibrosis in patients with severe aortic valve stenosis.

DETAILED DESCRIPTION:
AS is the most common valvular heart condition in the Western world. In response to increased afterload imposed by AS adaptive left ventricular (LV) remodelling occurs which in a course of a disease transitions from LV hypertrophy to maladaptive changes in the myocardium leading to cardiac decompensation and symptoms development. This transition is predominantly driven by myocardial fibrosis and myocyte cell death. Increasing evidence have demonstrated that presence of myocardial fibrosis, detected by cardiovascular magnetic resonance (CMR), could serve as an early marker of LV decompensation and predict adverse outcomes in patients with aortic stenosis. Currently, the indications for valvular replacement are based on the stenosis severity evaluated by echocardiography and the presence of symptoms.

The objective of the project is to identify parameters of non-invasive imaging modalities (two-dimensional echocardiography with an extended myocardial deformation analysis, 1.5 T CMR with T1 parametric map and late gadolinium enhancement (LGE) predictive of cardiac decompensation and to evaluate the prognostic significance of myocardial fibrotic changes in patients with severe degenerative AS. In patients with suspicion of cardiac amyloidosis, 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid (DPD) scintigraphy will be performed.

Study design: a prospective, open, case-driven, multicentre study (Lithuania, Denmark).

Investigators will assess LV structural and functional alterations before and 12 months after aortic valve intervention. Cardiac imaging data will be aligned with histopathological data from myocardial tissue samples collected at the time of aortic valve replacement in SAVR group. In patients with suspicion of cardiac amyloidosis, DPD scintigraphy and further evaluation regarding amyloidosis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (aortic valve area <1.0cm2 or aortic valve area index <0.6 cm2/m2
* Age ≥18 years.
* Signed informed patient consent form.

Exclusion Criteria:

* Severe valvular disease other than AS.
* Significant coronary heart disease requiring revascularisation.
* History of myocardial infarction.
* Previous cardiac surgery.
* Severe renal impairment eGFR <30ml/min/1.73m2.
* Any absolute contraindication to CMR.
* Inherited or acquired cardiomyopathy.
* Other medical conditions that limits life expectancy or precludes SAVR or TAVI.
* Pregnant or nursing women
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
* Patients in permanent atrial fibrillation.
* Significant chronic obstructive pulmonary disease (FEV1 <70% of predicted value)
* Patient with implanted devices (pacemaker, ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis without significant coronary artery disease (CAD), eligible for aortic valve intervention (SAVR or TAVI).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
A composite of all-cause mortality and MACE (Acute myocardial infarction, stroke, heart failure requiring hospitalisation) | 2 years

SECONDARY OUTCOMES:
Cardiovascular mortality | 2 years
Short term mortality | 30 days
  Intrahospital or 30 days mortality
Lengh of hospital stay | 30 days
Time to the event ( deathe of MACE) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sogaard, Prof., Principal Investigator — Aalborg University
Locations (2):
- Aalborg University Hospital, Aalborg, Denmark
- Vilnius University Hospital Santaros clinics, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balciunaite G, Palionis D, Zurauskas E, Skorniakov V, Janusauskas V, Zorinas A, Zaremba T, Valeviciene N, Aidietis A, Serpytis P, Rucinskas K, Sogaard P, Glaveckaite S. Prognostic value of myocardial fibrosis in severe aortic stenosis: study protocol for a prospective observational multi-center study (FIB-AS). BMC Cardiovasc Disord. 2020 Jun 8;20(1):275. doi: 10.1186/s12872-020-01552-8. PMID 32513178